CLINICAL TRIAL: NCT04817592
Title: Characterization of the Corneal Biomechanics of Patients Treated by Corneal Lenticule Extraction for Advanced Refractive Correction (CLEAR) to Correct Myopia
Acronym: CLEAR Biomech
Status: Not yet recruiting | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Basec Nr 2021-001-45
Record Dates: First submitted 2021-03-15; First posted 2021-03-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Myopia
Keywords: Cornea; SMILE; CLEAR
MeSH Terms: conditions — Myopia; Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Age1(20-25): The groups are divided as per age
  Interventions: Procedure: Corneal lenticule extraction for advanced refractive correction (CLEAR)
- Age2(25-30)
  Interventions: Procedure: Corneal lenticule extraction for advanced refractive correction (CLEAR)
- Age3(30-35)
  Interventions: Procedure: Corneal lenticule extraction for advanced refractive correction (CLEAR)
- Age4(35-40)
  Interventions: Procedure: Corneal lenticule extraction for advanced refractive correction (CLEAR)
- Age5(40-45)
  Interventions: Procedure: Corneal lenticule extraction for advanced refractive correction (CLEAR)

INTERVENTIONS:
Procedure: Corneal lenticule extraction for advanced refractive correction (CLEAR) — Routinely conducted procedure for correction of Myopia
  Other Names: SMILE

SUMMARY:
This study aims to perform biomechanical tests on extracted CLEAR lenticles that are routinely discarded after surgery. The investigators also aim to perform Brillouin microscopy to get an in-vivo assessment of the patient's cornea preoperatively and to correlate this data with the postoperative characterization of the extracted corneal lenticule. The characterization will be done with established biomechanical and morphologic tests.

DETAILED DESCRIPTION:
Refractive surgery techniques such as laser in situ keratomileusis (LASIK), corneal lenticule extraction (SMILE/CLEAR) and photorefractive keratectomy (PRK) are becoming increasingly popular among myopic patients. With current surgical planning tools, there is a reported 10-15 % chance of over/under correction, in particular with higher corrections. The biggest factor that leads to this discrepancy is the "one size fits all" approach. Patient specific characteristics of the eye such as the corneal material properties, are not considered in the surgical planning. This information is also essential for diagnosis and treatment of pathologies like keratoconus. New diagnostics devices based on e. g. Brillouin scattering are now introduced on the market, with the aim to provide an in-vivo quantification of the biomechanical tissue properties. However, the relationship between the Brillouin measurement and the biomechanical properties of the cornea is not fully understood yet. The investigators aim for determining an improved relationship between the optical Brillouin measurement performed in-vivo preoperatively and classical destructive biomechanical testing of the extracted corneal lenticule after the surgery. This lenticule is currently discarded after surgery.

The purpose of the study is to investigate the exact relationship between the classically determined material properties (by stress-/strain measurements) and optically obtained data by Brillouin scattering, which are collected during pre-op investigations. A precise characterization and relation between both measurements will allow clinicians to better predict surgical parameters and perform better refractive interventions. This information will also inform clinicians on the mechanical status of the cornea of patients suffering from subclinical keratoconus.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for CLEAR procedures for myopia (range: >-3D with an astigmatism <0.25D) in the age group 20-50 years.
* Willing and able to return for scheduled follow-up examinations
* Able to provide written informed consent and follow study instructions in English or German

Exclusion Criteria:

* Irregular corneal topo-/tomography (Asymmetry >1.0D within the inner 5mm)
* Previous intraocular or corneal surgery of any kind in the eye to be treated, including any type of surgery for either refractive or therapeutic purposes.
* History of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative intraocular pressure (IOP) > 21 mmHg in either eye.
* History of diabetes, diagnosed autoimmune disease, connective tissue disease or clinically significant atopic syndrome.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects voluntarily undergoing routinely prescribed CLEAR /SMILE intervention
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomechanics of extracted lenticule | 1 year
  During the CLEAR intervention, the lenticule extracted will be marked for physiological direction to identify the nasal-temporal and superior-inferior directions and stored at room temperature in normal culture medium from eye banking with 6% dextran. The mechanical experiments on these lenticules, will be performed within 24hours after extraction to preserve the sample properties. The samples will undergo uniaxial tensile testing in IROC using the UStretch (Cellscale, Waterloo, ON, Canada) device. Post tensile testing, the samples will be imaged using Second-harmonic imaging microscopy (SHG microscopy). SHG microscopy will be used to determine the in-plane probability distribution describing the orientation and density of the collagen fibrils present in the CLEAR lenticules. This information will be incorporated into a computational model which will simulate the uniaxial stress-strain measurements to further help us identify the parameters of a non-linear constitutive material model.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Büchler, Prof. Dr., Principal Investigator — University of Bern
Locations (1):
- IROC AG, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No